CLINICAL TRIAL: NCT04788953
Title: Clinical Trial of Solriamfetol for Excessive Sleepiness Related to Shift Work Disorder
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was stopped due to funding limitations.
Sponsor: Charles A. Czeisler, PhD, MD (Other)
Collaborators: Axsome Therapeutics, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Charles A. Czeisler, PhD, MD, Baldino Professor of Sleep Medicine, Division Chief, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-P-000509
Record Dates: First submitted 2021-03-02; First posted 2021-03-09 (Actual); Results first posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Excessive Sleepiness; Shift-work Disorder
Keywords: Excessive Daytime Sleepiness; Early Morning Shift Work
MeSH Terms: conditions — Disorders of Excessive Somnolence | interventions — solriamfetol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Solriamfetol (Sunosi) (Experimental): Participants will start at 75 mg and take that dose for 3 consecutive days. Participants will take their first 75mg dose on an early morning work day and take the next two 75 mg doses upon awakening regardless of their work schedule.
  They will then move to 150mg on the next early morning work day and for all subsequent early morning shift work days. The drug/placebo will be taken orally within 30 minutes after awakening, before the start of each early morning shift. Prior to the end of study of visit (Visit 5), drug will be taken at home within 30 minutes of awakening.
  Interventions: Drug: Solriamfetol Oral Tablet
- Control (Placebo Comparator): Participants randomized into the Control arm will receive a placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Solriamfetol Oral Tablet — The administered drug is SUNOSI (solriamfetol) tablets for oral use. Initial U.S. Approval: 2019
  Other Names: Sunosi
  Arms: Solriamfetol (Sunosi)
Drug: Placebo — Control subjects will receive placebo tablets for oral use.
  Arms: Control

SUMMARY:
In this research study the investigators want to learn more about whether the medication Solriamfetol improves daytime sleepiness in workers who start work at very early times (between 3 and 6am).

DETAILED DESCRIPTION:
Shift work has become increasingly common as the 24/7 global society has required more and more workers to do their jobs at irregular hours. According to the National Health Interview Survey in 2010, approximately 28.7% of the American workforce is engaged in work outside a regular day shift (outside 7 AM-to 6 PM). Working irregular hours poses a serious threat to the shift worker's physical, mental, and psychosocial health due to circadian misalignment and misplaced sleep. The most severe problems faced by shift workers are sleep disturbances and excessive sleepiness. The disruptions caused by shift work are recognized as a circadian rhythm sleep disorder in the International Classification of Sleep Disorders, 3rd Edition, and is called Shift Work Disorder [SWD]. SWD is characterized by excessive sleepiness (ES) during wakefulness, accompanied by a reduction of total sleep time and/or insomnia. Several studies have shown that 10-43% of shift workers are diagnosed with SWD, dependent on the criteria used.

Studies have shown that wake promoting agents can be used to treat ES in shift workers, ranging from caffeine to prescription pharmacological agents. Current Food and Drug Administration (FDA)-approved options for SWD patients with ES are modafinil and armodafinil. A three-month, double-blind trial of 209 randomized SWD patients showed that modafinil improves wakefulness and the ability to sustain attention working night shifts without negatively affecting daytime sleep. Furthermore, SWD patients who received modafinil had an improvement in clinical symptoms, reduced levels of sleepiness during night shift and during commute home, and proportionally fewer patients reported motor vehicle accidents or near accidents while commuting home. Czeisler and colleagues also performed a 12-week randomized, double-blind, placebo-controlled, parallel-group, multicenter study, which showed that armodafinil was well-tolerated and improved clinical conditions, wakefulness, attention and memory during night shifts in SWD patients without jeopardizing daytime sleep and reduced sleepiness during the commute home.

All these previous studies were described in SWD patients working night shifts, yet approximately 3 times as many individuals work shifts that start in the early morning compared with those who work night shifts. These early-morning shift workers are a unique, high-risk group because their early work start times (3:00 AM to 6:00 AM) require the workers to wake up in the middle of the night, close to their circadian nadir, resulting in curtailed sleep and commuting to work during times of high sleepiness. Previous research has shown that early-morning shift starts in particular are associated with increased sleepiness. To the investigators' knowledge, no studies have addressed the use of wake promoting agents for ES in early-morning shift workers.

In this clinical trial, the investigators will test whether Solriamfetol (SUNOSITM), a drug approved for the treatment of ES in patients with obstructive sleep apnea (OSA) and narcolepsy, is effective in: (1) decreasing sleepiness without reducing sleep duration or sleep quality; (2) improving work functioning; and (3) improving quality of life in early-morning shift workers diagnosed with ES associated with SWD.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women
2. Ages 18 to 64 years
3. Early-morning shift workers with a fixed work schedule (start times between 3 AM-6 AM, for at least 3 days per week)
4. ≥ 20 work hours per week, 6-hour to 12-hour shifts
5. ≥ 3-month history of working early morning shifts prior to the study
6. Shift work disorder (as measured by 4-item SWD screening questionnaire and SWD symptoms confirmed by clinician) with excessive sleepiness (as measured by the modified ESS) specifically related to early morning shifts
7. Baseline MWT average sleep latency <20 minutes on the first 4 scheduled naps
8. Body mass index 18.5 to 45 kg/m2
9. Normal thyroid stimulating hormone (TSH) level
10. Female participants must not be pregnant or breastfeeding.
11. Female participants must either be of non-childbearing potential or using a contraceptive method that is highly effective (with a failure rate of <1% per year), preferably with low user dependency, and agree to continue its use for at least 30 days after the last dose of study medication.
12. Male participants must agree to refrain from donating sperm and agree to remain abstinent from heterosexual intercourse or to use a male condom with female partners who are on an additional highly effective contraceptive method, both during the study and for at least 30 days after the last dose of study medication.
13. Are willing to refrain from any alcohol and nicotine-containing product use during the 24 hours prior to each MWT visit.
14. Are willing to refrain from any caffeine use on the day of the MWT visits.
15. Are willing and able to comply with the study requirements.

Exclusion Criteria:

1. History or presence of any acutely unstable medical condition, behavioral or psychiatric disorder, or surgical history that could affect the safety of the participant or interfere with study efficacy, safety, or the ability of the participant to complete the trial based on the judgment of the investigator.
2. Presence of renal impairment or calculated creatinine clearance < 60 mL/min.
3. Laboratory value(s) outside the laboratory reference range that is considered to be clinically significant by the investigator (clinical chemistry, hematology, and urinalysis; see Appendix II).
4. Hypothyroidism or hyperthyroidism, unless stabilized by appropriate medication for at least 3 months prior to screening.
5. Clinically significant EKG abnormality in the opinion of the investigator.
6. Presence of significant cardiovascular disease including but not limited to: myocardial infarction within the past year, unstable angina pectoris, symptomatic congestive heart failure (ACC/AHA stage C or D), revascularization procedures within the past year, uncontrolled atrial fibrillation, ventricular cardiac arrhythmias requiring automatic implantable cardioverter defibrillator or medication therapy, uncontrolled hypertension, systolic blood pressure ≥ 155 mmHg or diastolic blood pressure ≥ 95 mmHg (at Screening or Baseline), or any history of cardiovascular disease or any significant cardiovascular condition that in the investigator's opinion may jeopardize participant safety in the study.
7. History of bariatric surgery within the past year or a history of any gastric bypass procedure.
8. Use of an MAOI in the past 14 days or five half-lives (whichever is longer) prior to the Baseline Visit, or plans to use an MAOI during the study.
9. Pregnant or intention to become pregnant.
10. Breast-feeding or plans to breastfeed.
11. On long-term sick leave or with no history of work in the last 12 months
12. Diagnosis with sleep disorder (regardless of treatment status) other than SWD including: OSA, PLMD, other circadian rhythm sleep disorders, narcolepsy, or RLS determined by a previous sleep-lab diagnosis or during the home sleep test.
13. History of excessive caffeine use or anticipated excessive use (>600mg/day) during the study.
14. Use of any OTC or prescription medications that could affect the evaluation of EDS within a time period prior to the Baseline visit corresponding to at least 5 half-lives of the drug(s) or planned use of such drug(s) at some point throughout the duration of the treatment period. Examples of excluded medications include OTC sleep aids, stimulants (e.g. methylphenidate, amphetamines, modafinil, and armodafinil), sodium oxybate, pemoline, pitolisant, bupropion, trazodone, vortioxetine, duloxetine, tricyclic antidepressants, hypnotics, benzodiazepines, barbiturates, and opioids.
15. Received an investigational drug in the past 30 days or 5 half-lives (whichever is longer) prior to the Baseline visit or plans to use an investigational drug (other than the study drug) during the study.
16. History or presence of bipolar disorder, bipolar-related disorders, schizophrenia, schizophrenia spectrum disorders, or other psychotic disorders according to DSM-5 criteria.
17. Current or recent (within the past 2 years) diagnosis of a moderate or severe substance use disorder (excluding caffeine) according to DSM-5 criteria. Nicotine use disorder is exclusionary only if it has an effect on sleep (i.e., a participant who routinely awakens at night to smoke) or will interfere with study compliance.
18. Current, recent (within the past 2 years), or seeking treatment for a substance-related disorder.
19. Positive urine drug screen (UDS) for opiates, phencyclidine (PCP), cocaine, cannabinoid (THC), or amphetamines at Screening or at any point throughout the duration of the study, except for a prescribed drug (e.g., amphetamine) at Screening.
20. History of regular heavy use of tetrahydrocannabinol containing products. Recreational users of cannabis may be repeat UDS tested once during the Screening period. If this is negative, the participant may be allowed to enter the study.
21. Positive alcohol test at Screening. Binge drinking (5 or more drinks per day for men, 4 or more drinks per day for women) within the past month.
22. History of PKU or history of hypersensitivity to phenylalanine-derived products.
23. Previous exposure to solriamfetol (JZP-110, ADX-N05, R228060, or YKP-10A).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2024-04-06 (Actual); Study Completion 2024-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles A Czeisler, PhD,MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Zitting KM, Gilmore KR, Lockyer BJ, Leary EB, Wang W, Issa NC, Quan SF, Williams JS, Duffy JF, Czeisler CA. Solriamfetol for Excessive Sleepiness in Early-Morning Shift Work Disorder. NEJM Evid. 2026 Feb;5(2):EVIDoa2500190. doi: 10.1056/EVIDoa2500190. Epub 2026 Jan 27. PMID 41590992

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via online advertisements, radio advertisements and fliers between July 2021 and April 2024.
Pre-assignment Details: 84 participants were enrolled in the study. Of these 84 participants, 6 were excluded before assigment (5 due to changes in participants' work schedules making them ineligible and 1 because the study was terminated/stopped study early). A total of 78 participants started taking solriamfetol or placebo.
Period: Overall Study
Arm/Group | Solriamfetol (Sunosi) | Control
Started | 40 | 38
Completed | 38 | 36
Not Completed | 2 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Data were analyzed for all participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Solriamfetol (Sunosi) | Control | Total
Number analyzed (Participants) | 38 | 36 | 74
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 40 [28 to 45] | 34 [28 to 48] | 37 [28 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 25 | 22 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 5 | 16
  Not Hispanic or Latino | 26 | 27 | 53
  Unknown or Not Reported | 1 | 4 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 2 | 6
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 25 | 23 | 48
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 1 | 5 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38 | 36 | 74
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m2] | 27 [24 to 35] | 29 [24 to 33] | 28 [24 to 33]

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Sleep Latency
Description: Sleep latency was assessed with a Maintenance Wakefulness Test (MWT) at Visit 2 (Baseline) and again at Visit 5 (End-of-Treatment). The MWT started ~2 hours after participant's usual wake time and consisted of four 40-minute trials (2, 4, 6, and 8 hours after usual wake time). Participants were fitted with polysomnography (PSG) and instructed to stay awake. Each trial was monitored and the trial was ended after PSG-sleep occurred or after 40 minutes if no sleep occurred. Sleep latency (in minutes) was calculated as the time between trial start time and sleep onset time. Change in mean sleep latency (i.e., averaged sleep latency across the four trials) from Visit 2 to Visit 5 was calculated for each participant.
Time Frame: Study Visit 2 (i.e., Baseline Visit) and Study Visit 5 (i.e., End-of-Treatment Visit after 4 weeks on solriamfetol or placebo)
Population: Data were analyzed for all participants who completed the study.
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Solriamfetol (Sunosi) | Control
Number analyzed (Participants) | 38 | 36
minutes | 12.6 [10.0 to 15.2] | 3.2 [0.6 to 5.8]
Statistical Analysis 1: Comparison: Solriamfetol (Sunosi) vs Control; The statistical null hypothesis was that solriamfetol does not improve change in MWT scores versus placebo after 4 weeks of treatment (H0: µsol - µpl ≤ 0). Study was designed to have 97% power to detect a difference of 5.7 minutes or greater on MWT sleep latency (α=0.05, assumed σ=7.2) with 100 participants. Blinded interim power analysis on the baseline data conducted in October 2023 indicated the trial would have >99% power to detect a similar difference with only 74 participants; Test type: Superiority; p < 0.001, Mixed Models Analysis — Change from baseline using mixed-effects tobit regression model (censored normal). Group (Solriamfetol, Placebo), visit (Baseline, End-of-Treatment), trial (1-4) main factors and their interactions. Covariates considered: age, sex, ethnicity, race; P-value is difference between groups

2. Secondary Outcome: Change in Karolinska Sleepiness Scale Score
Description: Subjective sleepiness was assessed with a Karolinska Sleepiness Scale (KSS, Åkerstedt & Gillberg, 1990). The KSS was administered to the participant ~5 minutes before the start of each four MWT trial at Visit 5 (Baseline) and again at Visit 5 (End-of-Treatment). The KSS scores range from 1 (very alert) to 9 (very sleepy), with higher scores indicating higher levels of sleepiness. Change in the mean KSS score (i.e., averaged score across the four trials) from Visit 2 to Visit 5 was calculated for each participant.
Time Frame: as for outcome 1
Population: Data were analyzed for all participants who completed the study.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Solriamfetol (Sunosi) | Control
Number analyzed (Participants) | 38 | 36
score on a scale | -1.7 [-2.0 to -1.3] | -0.5 [-0.8 to -0.1]
Statistical Analysis 1: Comparison: Solriamfetol (Sunosi) vs Control; Test type: Superiority; p < 0.001, Mixed Models Analysis — Change from baseline using mixed-effects linear regression model. Group (Solriamfetol, Placebo), visit (Baseline, End-of-Treatment), trial (1-4) main factors and their interactions. Covariates considered: age, sex, ethnicity, race; P-value is difference between groups

3. Secondary Outcome: Change in Clinician's Global Impression of Change Score
Description: Overall change in participant's clinical condition was assessed with a Clinician's Global Impression of Change scale (CGI-Change, Guy, 1976). The CGI-change was conducted at Visit 5 (End-of-Treatment) by a study doctor who rated the participant. The scores range from 1 (very much improved) to 7 (very much worse), with lower scores indicating improved condition. Data were dichotomized such that scores 1-3 (very much improved, much improved, minimally improved) were considered to indicate improvement and scores 4-7 (no change, minimally worse, much worse, very much worse) were considered to indicate no improvement. Improvement was calculate as the percentage of participants in each group who reported improved scores.
Time Frame: Study Visit 5 (i.e., End-of-Treatment Visit after 4 weeks on solriamfetol or placebo)
Population: Data were analyzed for all participants who completed the study. CGI-C data for 2 patients in the Solriamfetol Group and 1 patient in the Placebo Group was lost due to technical error.
Measure: Number; unit: percent of improved participants
Arm/Group | Solriamfetol (Sunosi) | Control
Number analyzed (Participants) | 36 | 35
percent of improved participants | 77.8 | 48.6
Statistical Analysis 1: Comparison: Solriamfetol (Sunosi) vs Control; Test type: Superiority; p = 0.01, Chi-squared — Chi-squared tests performed on dichotomized CGI-Change data ("Improved" [very much improved, much improved, minimally improved] vs. "Not Improved" [no change, minimally worse, much worse, very much worse]); P-value is difference between groups

4. Secondary Outcome: Change in Patient's Global Impression of Change Score
Description: Participant's overall perception of change in their condition (i.e., excessive sleepiness) was assessed with a Patient's Global Impression of Change scale (PGI-Change, Guy, 1976). The PGI-C was administered to the participant at Visit 5 (End-of-Treatment). The scores ranged from 1 (no change or worse) to 7 (a great deal better), with higher scores indicating improved condition. Data were dichotomized such that scores 1-2 (no change or worse, hardly any change) were considered to indicate no improvement, and scores 3-7 (a little better, somewhat better, moderately better, better, a great deal better) were considered to indicate improvement.
Time Frame: Study Visit 5 (i.e., End-of-Treatment Visit after 4 weeks on solriamfetol or placebo)
Population: Data were analyzed for all participants who completed the study.
Measure: Number; unit: percent of improved participants
Arm/Group | Solriamfetol (Sunosi) | Control
Number analyzed (Participants) | 38 | 36
percent of improved participants | 78.9 | 47.2

5. Other Pre Specified Outcome: Change in Overall Work Impairment Score From the Work Productivity and Activity Impairment Questionnaire
Description: Work impairment was assessed with a Work Productivity and Activity Impairment-Specific Health Problem questionnaire (WPAI-SHP, Reilly et al., 1993; Emsellem et al., 2020), with excessive sleepiness as the specific health problem. The WPAI-SHP questionnaire was administered to the participant at Visit 2 (Baseline) and again at Visit 5 (End-of-Treatment). Overall work impairment score, which ranges from 0 to 100 with higher score indicating more impairment, was calculated from the WPAI-SHP subscales according to the WPAI scoring manual by Dr. Reilly. Change in the overall work impairment score from Visit 2 to Visit 5 was calculated for each participant.
Time Frame: as for outcome 1
Population: Data were analyzed for all participants who completed the study.
Measure: Least Squares Mean (95% Confidence Interval); unit: overall work impairment score
Arm/Group | Solriamfetol (Sunosi) | Control
Number analyzed (Participants) | 38 | 36
overall work impairment score | -21.6 [-31.5 to -11.7] | -4.9 [-15.0 to 5.3]
Statistical Analysis 1: Comparison: Solriamfetol (Sunosi) vs Control; Test type: Superiority — Change from baseline using mixed-effects linear regression model. Group (Solriamfetol vs. Placebo) and visit (Baseline vs. End-of-Treatment) as main factors and their interactions. Covariates considered: age, sex, ethnicity, race; p = 0.02, Mixed Models Analysis; P-value is difference between groups

6. Other Pre Specified Outcome: Change in Functional Outcomes of Sleep Questionnaire Score
Description: Subjective global functioning was assessed with the short version of the Functional Outcomes of Sleep Questionnaire (FOSQ-10; Chasens et al., 2009). The FOSQ-10 was administered to the participant at Visit 2 (Baseline) and again at Visit 5 (End-of-Treatment). The FOSQ-10 consists of ten subscales with each subscale ranging from 1 (extreme difficulty) to 4 (no difficulty). The FOSQ-10 total score, which was calculated as the mean-weighted item score computed from the ten subscales, ranges from 5 to 20 with higher scores indicating less functional impairment. Change in FOSQ-10 total score from Visit 2 to Visit 5 was calculated for each participant.
Time Frame: as for outcome 1
Population: Data were analyzed for all participants who completed the study.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Solriamfetol (Sunosi) | Control
Number analyzed (Participants) | 38 | 36
score on a scale | 2.0 [0.9 to 3.0] | 1.6 [0.5 to 2.7]
Statistical Analysis 1: Comparison: Solriamfetol (Sunosi) vs Control; Test type: Superiority; p = 0.64, Mixed Models Analysis — Change from baseline using mixed-effects linear regression model. Group (Solriamfetol vs. Placebo) and visit (Baseline vs. End-of-Treatment) as main factors and their interactions. Covariates considered: age, sex, ethnicity, race; P-value is difference between groups

7. Other Pre Specified Outcome: Change in Sheehan Disability Scale Score
Description: The impact of excessive sleepiness on subjective global functioning was assessed with a Sheehan Disability Scale (SDS; Sheehan & Sheehan, 2008). The questionnaire was administered to the participants at Visit 2 (Baseline) and again at Visit 5 (End-of-Treatment). The SDS consists of five subscales, with the scores for the three subscales (work, social, and family life) that are used for calculating the total score ranging from 0 (not at all impacted) to 10 (extremely impacted). The SDS total score, which was calculated as the sum of the three subscale scores, ranges from 0 to 30 with higher scores indicating greater functional impairment. Change in the SDS total score from Visit 2 to Visit 5 was calculated for each participant.
  which ranges from 0 to 30,
Time Frame: as for outcome 1
Population: Study Visit 2 (i.e., Baseline Visit) and Study Visit 5 (i.e., End-of-Treatment Visit after 4 weeks on solriamfetol or placebo)
Measure: Least Squares Mean (95% Confidence Interval); unit: total score on a scale
Arm/Group | Solriamfetol (Sunosi) | Control
Number analyzed (Participants) | 38 | 36
total score on a scale | -6.8 [-9.3 to -4.4] | -3.1 [-5.6 to -0.6]
Statistical Analysis 1: Comparison: Solriamfetol (Sunosi) vs Control; Test type: Superiority; p = 0.04, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; P-value is difference between groups

8. Other Pre Specified Outcome: Change in Total Sleep Time
Description: Total Sleep Time (TST) was assessed with actigraphy. Participants wore a wrist activity monitor throughout the study (i.e., 2 weeks of baseline and 4 weeks of treatment). The actigraphy data from the main sleep periods were manually scored in 30-second epochs, and TST was calculated in minutes for each study day. Change in TST from baseline to treatment was calculated for each participant.
Time Frame: Baseline Segment (2 weeks) and Treatment Segment (4 weeks)
Population: Data were analyzed for all participants who completed the study over the 4 week treatment period. Actigraphy data for the last 2 weeks of treatment were missed for 1 patient in the Solriamfetol Group due to a damaged wrist activity monitor and for 1 patient in the Placebo Group due to technical failure.
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes
Arm/Group | Solriamfetol (Sunosi) | Control
Number analyzed (Participants) | 38 | 36
minutes | -3.6 [-13.5 to 6.3] | -7.2 [-17.3 to 2.9]
Statistical Analysis 1: Comparison: Solriamfetol (Sunosi) vs Control; Test type: Superiority; p = 0.61, Mixed Models Analysis — Change from baseline using mixed-effects linear regression model. Group (Solriamfetol vs. Placebo) and Condition (Baseline vs. Treatment) as main factors and their interactions. Covariates considered: age, sex, ethnicity, race; P-value is difference between groups

9. Other Pre Specified Outcome: Change in Sleep Fragmentation Index
Description: Sleep disturbances were assessed with actigraphy-derived fragmentation index. Participants wore a wrist activity monitor throughout the study (i.e., 2 weeks of baseline and 4 weeks of treatment). The actigraphy data from the main sleep periods were manually scored in 30-second epochs in the MotioWare software (CamNtech, Cambridge, UK). MotionWare defines the fragmentation index as the sum of the percentages of mobile time and immobile bouts immobile bouts below or equal to 1 minute during the sleep period, which is a unitless measure. Change in fragmentation index from baseline to treatment was calculated for each participant.
Time Frame: Baseline Segment (2 Weeks) and Treatment Segment (4 Weeks)
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: unitless measure
Arm/Group | Solriamfetol (Sunosi) | Control
Number analyzed (Participants) | 38 | 36
unitless measure | 0.5 [-0.5 to 1.5] | 0.9 [-0.1 to 1.9]
Statistical Analysis 1: Comparison: Solriamfetol (Sunosi) vs Control; Test type: Superiority; p = 0.57, Mixed Models Analysis — [p-value comment as in outcome 8, analysis 1]; P-value is difference between groups

10. Other Pre Specified Outcome: Change in Epworth Sleepiness Scale Score
Description: Subjective sleepiness was assessed with a modified Epworth Sleepiness Scale (ESS, Johns, 1990, 1997). The ESS was administered to the participant at Visit 2 (Baseline) and again at Visit 5 (End-of-Treatment). The ESS consists of eight subscales with each subscale ranging from 0 (never doze) to 3 (high change to doze off). The ESS total score, which was calculated as the sum of the eight subscalescores, ranges from 0 (normal levels of sleepiness) to 24 (severe excessive sleepiness) with higher scores indcating higher levels of sleepiness. Change in the ESS total score from Visit 2 to Visit 5 was calculated for each participant.
  total score, which ranges from 0 to 24 (0=normal level of sleepiness, 24=severe excessive sleepiness), was calculated by summing the scores from the eight subscales. Change in ESS total score from Visit 2 to Visit 5 was calculated for each participant.
Time Frame: Study Visit 2 (i.e., Baseline Visit) and Study Visit 5 (i.e., End of Treatment Visit after 4 weeks on solriamfetol or placebo)
Population: Data were analyzed for all participants who completed the study.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Solriamfetol (Sunosi) | Control
Number analyzed (Participants) | 38 | 36
score on a scale | -7.2 [-8.8 to -5.5] | -2.4 [-4.1 to -0.8]
Statistical Analysis 1: Comparison: Solriamfetol (Sunosi) vs Control; Test type: Superiority; p < 0.001, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; P-value is difference between groups

ADVERSE EVENTS:
Time Frame: Adverse events data for each participant was collected for approximately 4 weeks. This spanned the time period between Visit 3 (solriamfetol/placebo dispensed to the participant) and Visit 5 (last solriamfetol/placebo dose).
Description: Adverse events were collected from participant reports during study visits, scheduled check-ins, and other interactions with the participants. Adverse event reporting includes all adverse events that occurred between study visits 3 and 5 for participants who took at least one dose of drug/placebo.
Groups:
- Solriamfetol (Sunosi): Participants will start at 75 mg and take that dose for 3 consecutive days. Participants will take their first 75mg dose on an early morning work day and take the next two 75 mg doses upon awakening regardless of their work schedule.
  They will then move to 150mg on the next early morning work day and for all subsequent early morning shift work days. The drug/placebo will be taken orally within 30 minutes after awakening, before the start of each early morning shift. Prior to the end of study of visit (Visit 5), drug will be taken at home within 30 minutes of awakening.
  Solriamfetol Oral Tablet: The administered drug is SUNOSI (solriamfetol) tablets for oral use. Initial U.S. Approval: 2019
Arm/Group | Solriamfetol (Sunosi) | Control
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/38
Other Adverse Events (participants affected / at risk) | 40/40 | 35/38
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Solriamfetol (Sunosi) (N=40) | Control (N=38)
abnormal dreams (General disorders) | 3 | 0
anxiety (Psychiatric disorders) | 3 | 0
arrhythmias (Cardiac disorders) | 0 | 2
cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
covid-19 (Respiratory, thoracic and mediastinal disorders) | 1 | 2
decreased appetite (Metabolism and nutrition disorders) | 4 | 0
diarrhea (Gastrointestinal disorders) | 2 | 1
dizziness (Nervous system disorders) | 3 | 2
feeling jittery (General disorders) | 4 | 2
headache (Nervous system disorders) | 12 | 10
insomnia (Psychiatric disorders) | 1 | 2
lethargy (General disorders) | 1 | 3
nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
nausea (Gastrointestinal disorders) | 7 | 5
sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-16): https://cdn.clinicaltrials.gov/large-docs/53/NCT04788953/Prot_SAP_000.pdf
  • Informed Consent Form (2025-01-13): https://cdn.clinicaltrials.gov/large-docs/53/NCT04788953/ICF_001.pdf